CLINICAL TRIAL: NCT05426590
Title: Evaluation of Corneal Endothelial Changes After Uneventful Phacoemulsification in Diabetic and Non-diabetic Patients in Relation to the Level of Glcosylated Hemoglobin Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marwa Ahmed (Other)
Responsible Party: Sponsor-Investigator, Marwa Ahmed, Clinical professor, Cairo University
Organization: Cairo University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KasrAlAiny
Record Dates: First submitted 2022-06-04; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Corneal Endothelial Changes After Phacoemulsification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic patient (Active Comparator): Patient with diabetes will undergo cataract surgery
  Interventions: Device: Specular biomicroscopy
- Non diabetic patients (Active Comparator): Healthy non diabetic patients will undergo cataract surgery
  Interventions: Device: Specular biomicroscopy

INTERVENTIONS:
Device: Specular biomicroscopy — Specular microscopy will be done before and 3 weeks after cataract surgery

SUMMARY:
Evaluation of corneal endothelial changes after uneventful phacoemulsification in diabetic and non-diabetic patients using specular biomicroscopy in relation to the level of glcosylated hemoglobin level

DETAILED DESCRIPTION:
86 patients will be divided into two equal groups of diabetic and non-diabetic patients will undergo phacoemulsification of cataract will be evaluated thier endocelium before surgery and 3 weeks after surgery to detect the effect of level of glcosylated hemoglobin on the endothelial changes after uneventful phacoemulsification

ELIGIBILITY:
Inclusion Criteria:

* Diabetics and non-diabetic patients undergo cataract surgery
* Age between 50-60 years old
* Corrected distance visual acuity<0.4
* Gender: both genders.

Exclusion Criteria:

* Chronic Ocular diseases (glaucoma,uveitis, amblyopia, strabismus,keratoconus, corneal opacity).
* corneal dystrophy History of previous keratitis or viral corneal infection. Corneal dystrophy Ocular trauma. Previous ocular surgery. Complicated cataract surgery

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-11-17 (Estimated); Study Completion 2022-11-17 (Estimated)

PRIMARY OUTCOMES:
Defferentiate patients into diabetic and non-diabetic patients according to the endothelial changes after uneventful phacoemulsification | 6 monthes
  Detect effect of glycosylated hemoglobin level after uneventful phacoemulsification in diabetic and non-diabetic patients

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hosny, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt